CLINICAL TRIAL: NCT01577797
Title: A Cognitive Behavioral Therapy-Based Text Messaging Intervention for Methamphetamine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Leaf Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-1
Record Dates: First submitted 2012-04-05; First posted 2012-04-16 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine; Drug Abuse; Substance Abuse; Amphetamine; Dependence; Addiction; Craving; Cognitive Behavioral Therapy; Text Messaging
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-based text messages - Week 1 or 3 (Experimental): One week CBT-based text messages followed by a 1-week washout period (Week 2)
  Interventions: Behavioral: Text messages
- Placebo text messages - Week 3 or 1 (Placebo Comparator)
  Interventions: Behavioral: Text messages

INTERVENTIONS:
Behavioral: Text messages — Messages sent at random intervals 4 times per day during weeks 1 and 3. Subjects can also request messages if they are craving methamphetamine

SUMMARY:
This Phase I, randomized, 22-day crossover study seeks to improve treatment outcomes for methamphetamine-dependent subjects by developing a cognitive behavioral therapy (CBT)- based short message service (SMS) text messaging intervention as an adjunct to CBT group therapy.

DETAILED DESCRIPTION:
Psychosocial therapies for methamphetamine (MA) addiction all have limited effectiveness, and patients treated for MA dependence have a high rate of relapse. Additionally, there are no currently approved medications for MA dependence. Thus, a significant need exists for add-on therapy for treatment of MA addiction. CBT-based text messaging could serve as a real-time intervention when craving and risk of MA use are high and patients are not in the clinic. It could further serve to reinforce CBT group therapy. If found efficacious, fully-automated CBT-based text messaging would be a relatively inexpensive adjunctive therapy that could be readily scaled up for use in a large number of patients. Additionally, this type of text messaging intervention also could be tailored to individual users, which may enhance its efficacy. This Phase I randomized crossover study will evaluate the feasibility and preliminary efficacy of CBT-based text messages in conjunction with CBT group therapy delivered over a 22-day period in MA users in the San Francisco Bay Area.

ELIGIBILITY:
Main inclusion criterion:

* English-speaking adults who are currently seeking treatment for methamphetamine addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention in methamphetamine users | 22 days
  Subjects will respond to >50% of text messaging inquiries (about the usefulness of the messages, maximum degree of craving, and whether they have used that day).

SECONDARY OUTCOMES:
Acceptability of the intervention in methamphetamine users | 22 days
  Based on responses to follow-up visit questionnaires, is 4 times per day the "right amount" of text messages for subjects to receive each day? Is a 13-hour period in which subjects would receive messages appropriate? Was the software system selected for this study acceptable? Were the CBT-based text messages overall perceived as useful? Were the placebo text messages overall perceived as useful?

CONTACTS AND LOCATIONS:
Overall Officials: S. Alex Stalcup, MD, Principal Investigator — New Leaf Treatment Center
Locations (1):
- New Leaf Treatment Center, Lafayette, California, United States